CLINICAL TRIAL: NCT00285714
Title: An Analysis of the Clinical Applicability of a Three-Dimensional Imaging Platform Used to Register the Influence of Orthognathic Surgery on Facial Hard and Soft Tissue in Patients With Congenital Maxillofacial Deformities.
Brief Title: 3D Imaging of Hard and Soft Tissue in Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3D_MKC590_JP01
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2007-07-27 (Estimated); Status verified 2007-07

CONDITIONS: Craniofacial Abnormalities; Maxillofacial Abnormalities; Cleft Lip; Cleft Palate
Keywords: 3D computer assisted imaging; maxillofacial surgery; cephalometry; normative value
MeSH Terms: conditions — Craniofacial Abnormalities; Maxillofacial Abnormalities; Cleft Lip; Cleft Palate

INTERVENTIONS:
Procedure: 3D stereophotogrammetric imaging
Procedure: 3D CT-imaging with cone-beam CT
Procedure: Case report form

SUMMARY:
The primary objective of this clinical trial is to assess the influence of orthognathic surgery on facial soft tissue, such as changes (volume, linear, angular) of facial hard and soft tissue, in three dimensions, so enabling the setup of 3D normative value tables.

ELIGIBILITY:
Inclusion Criteria:

* Dysgnathic deformity
* Caucasian
* > 15 years
* No history of orthognathic surgery
* Informed Consent

Exclusion Criteria:

* < 15 years
* History of Orthognathic surgery
* Not Caucasian

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-02; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
All changes (volumetric, linear or angular) of facial hard and soft tissue caused by orthognathic surgery at 1 months, 6 months, 12 months and 24 months.

SECONDARY OUTCOMES:
All postoperative changes in functionality at 1 year
patients' satisfaction of facial proportions at 1 year
surgeons' satisfaction of the 3D planning platform at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan J Bergé, Prof, MD, DMD, PhD,, Study Director — Radboud University Medical Center; Filip AC Schutyser, MsC, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Hospital Gelderse Vallei, Ede
  - Radboud University Nijmegen Medical Centre, Nijmegen